CLINICAL TRIAL: NCT05327075
Title: Premenstrual Dysphoric Disorder:Knowledge,Attitude and Practice Among Egyptian Females.Results of Surveying Two Centers in Delta Region
Brief Title: Premenstrual Dysphoric Disorder:Knowledge,Attitude and Practice Among Egyptian Females
Acronym: PMDD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Eman Ibrahim Abd Elrehim, Lecturer in Department of obstetrics and gynecology, Damietta Faculty of Medicine, Al-Azhar University, Al-Azhar University
Other Study IDs: IRB 00012367-22-03-001
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Premenstrual Dysphoric Disorder
MeSH Terms: conditions — Premenstrual Dysphoric Disorder | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — it is in the form of questionnaire and scoring tool

SUMMARY:
it is a cross-sectional study conducted in female patients attending outpatient clinc in our university hospital to assess their awareness regarding the symptoms of premenstrual dysphoric disorders.

DETAILED DESCRIPTION:
this study will be conducted on females in the reproductive age attending the gynecological outpatient clinic to assess the prevalence of premenstrual dysphoric disorder(eeiPMDD) and their awareness regarding the symptoms of PMDD and the impact of these symptoms on their quality of life using questionnaire including ( knowledge , attitude and practice) of those Egyptian females.

ELIGIBILITY:
Inclusion Criteria:

females in reproductive age

history of regular menstruation

Exclusion Criteria:

history of any psychological disorders

history of chemotherapy in last 6 months

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — the participants in this study including females in reproductive age
Study Population: the study will include females attending gynecological clinics in two hospitals in delta region
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
questionnaire " awareness of participants regarding PMDD symptoms" | during the study, an avarege 1 month
  knowledge , attitude and practice through the time of questionnaire

SECONDARY OUTCOMES:
questionnaire "impact of the PMDD symptoms on the participants life" | 3 months
  impact on their life questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar University Hospital in Damietta, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided